CLINICAL TRIAL: NCT04498052
Title: Evaluation of a Scalable Decision Support and Shared Decision Making Tool for Lung Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kensaku Kawamoto, MD, PhD, MHS, Associate Chief Medical Information Officer, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UUtah_00125797
Record Dates: First submitted 2020-07-17; First posted 2020-08-04 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Early Detection of Cancer; Lung Neoplasms
Keywords: Lung Cancer Screening; Clinical Decision Support; Shared Decision Making
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: interrupted time series
Masking Description: no masking due to the nature of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients eligible for LDCT lung cancer screening (Experimental): This population will consist of patients eligible for, or potentially eligible for, LDCT lung cancer screening according to 2013 USPSTF guidelines. The inclusion criteria are (i) >= 55 years and <= 80 years old at the time of the visit; (ii) does not already have lung cancer; and (iii) meets USPSTF smoking criteria for LDCT screening (30+ pack-year smoking history and current smoker or quit in the past 15 years) or may meet the criteria if a complete smoking history were taken.
  Interventions: Other: EHR-integrated Shared Decision Making Tool and Clinical Decision Support for Lung Cancer Screening

INTERVENTIONS:
Other: EHR-integrated Shared Decision Making Tool and Clinical Decision Support for Lung Cancer Screening — The intervention will consist of the following core items:
  In period 1:
  * An EHR-integrated shared decision making (SDM) tool for providing information on the risks and benefits of lung cancer screening through low-dose computed tomography (LDCT) testing. This intervention is referred to as Decision Precision+.
  * Suggestions in the EHR to offer SDM for LDCT for patients eligible for lung cancer screening according to USPSTF guidelines. These suggestions include those provided by the EHR's "Health Maintenance" module as well as an EHR-integrated "Disease Manager" system for disease management and health maintenance.
  In period 2:
  - Same as period 1 + simple patient reminders in the patient portal.
  Following roll-out, clinic leaders may also receive periodic feedback on use of the intervention and LDCT screening rates, as well as advice on how to improve intervention adoption.

SUMMARY:
The purpose of this project is to increase appropriate low-dose computed tomography (LDCT) lung cancer screening through the development and wide dissemination of patient-centered clinical decision support (CDS) tools that (1) are integrated with the electronic health record (EHR) and clinical workflows, (2) prompt for shared decision making (SDM) when patients meet screening criteria, and (3) enable effective SDM using individually-tailored information on the potential benefits and harms of screening. The study will promote standard of care that is endorsed by the Centers for Medicare & Medicaid Services (CMS) and the US Preventive Services Task Force (USPSTF).

DETAILED DESCRIPTION:
The purpose of this project is to increase appropriate low-dose computed tomography (LDCT) lung cancer screening through the development and wide dissemination of patient-centered clinical decision support (CDS) tools that (1) are integrated with the electronic health record (EHR) and clinical workflows, (2) prompt for shared decision making (SDM) when patients meet screening criteria, and (3) enable effective SDM using individually-tailored information on the potential benefits and harms of screening. The study will promote standard of care that is endorsed by the Centers for Medicare & Medicaid Services (CMS) and the US Preventive Services Task Force (USPSTF). This project is supported both operationally and by an Agency for Healthcare Research and Quality (AHRQ) R18 grant.

This project will leverage Decision Precision, a validated Web-based tool for LDCT SDM developed at the Veterans Health Administration, as well as an initial version of Decision Precision+, an EHR-integrated version of the tool which can be accessed directly in the EHR and auto-populate relevant patient data in the tool instead of requiring manual data entry.

This study will be an 18-month interrupted time series study conducted at the University of Utah Health primary care clinics.

ELIGIBILITY:
Inclusion Criteria:

* receives care at University of Utah primary care clinics;
* does not already have lung cancer;
* meets USPSTF criteria for LDCT screening (currently, age >= 55 years and <= 80 years old at the time of the visit; 30+ pack-year smoking history and current smoker or quit in the past 15 years).

Exclusion Criteria:

* None

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1855 (Actual)
Dates: Start 2020-08-23 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2024-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kensaku Kawamoto, MD, PhD, MHS, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
We are not planning to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Tammemagi MC, Katki HA, Hocking WG, Church TR, Caporaso N, Kvale PA, Chaturvedi AK, Silvestri GA, Riley TL, Commins J, Berg CD. Selection criteria for lung-cancer screening. N Engl J Med. 2013 Feb 21;368(8):728-36. doi: 10.1056/NEJMoa1211776. PMID 23425165
- [Derived] Kukhareva PV, Li H, Caverly TJ, Fagerlin A, Del Fiol G, Hess R, Zhang Y, Butler JM, Schlechter C, Flynn MC, Reddy C, Choi J, Balbin C, Warner IA, Warner PB, Nanjo C, Kawamoto K. Lung Cancer Screening Before and After a Multifaceted Electronic Health Record Intervention: A Nonrandomized Controlled Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2415383. doi: 10.1001/jamanetworkopen.2024.15383. PMID 38848065
- [Derived] Kukhareva PV, Li H, Caverly TJ, Del Fiol G, Fagerlin A, Butler JM, Hess R, Zhang Y, Taft T, Flynn MC, Reddy C, Martin DK, Warner IA, Rodriguez-Loya S, Warner PB, Kawamoto K. Implementation of Lung Cancer Screening in Primary Care and Pulmonary Clinics: Pragmatic Clinical Trial of Electronic Health Record-Integrated Everyday Shared Decision-Making Tool and Clinician-Facing Prompts. Chest. 2023 Nov;164(5):1325-1338. doi: 10.1016/j.chest.2023.04.040. Epub 2023 May 3. PMID 37142092

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a non-randomized control study, where all eligible patients who had a visit in a pre-specified time period were assigned to that period. Therefore, some patients in periods 1 and 2 were the same, but some were different, resulting in 1855 patients in total, including 1104 in the baseline period, 1219 patients in period 1, and 1255 patients in period 2.
Period: Period 1 (Clinician-facing Intervention)
Arm/Group | Patients Eligible for LDCT Lung Cancer Screening
Started | 1219
Completed | 1219
Not Completed | 0
Period: Period 2 (Clinician + Patient Tools)
Arm/Group | Patients Eligible for LDCT Lung Cancer Screening
Started | 1255
Completed | 1255
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants: Study eligibility criteria were evaluated at the level of primary care visits (office visits or telehealth visits) during the study period. Patients were eligible if they met 2013 USPSTF LCS eligibility criteria at the time of the visit and had at least 1 primary care visit in the preceding year. Per USPSTF guidelines, a person qualified for LCS if they were aged 55 to 80 years, had a smoking history of 30 pack-years or greater, actively smoked or had quit in the previous 15 years, and had not been diagnosed with lung cancer.
Arm/Group | Participants
Number analyzed (Participants) | 1104
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65.0 [60.8 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 470
  Male | 634
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American, non-Hispanic | 20
  Hispanic, any race | 59
  White, non-Hispanic | 946
  Other | 79
Region of Enrollment [Number; unit: participants]
  United States | 1104
No. visits per patient [Median (Inter-Quartile Range); unit: visits] | 3.0 [1.0 to 5.0]
High-benefit personalized screening benefit level [Count of Participants; unit: Participants] — The screening benefit level was reported in accordance with guidance from the American College of Chest Physicians to identify patients who might obtain the most benefit from screening (high-benefit patients). To identify high-benefit patients, we used LYFS-CT models, with a benchmark of an anticipated gain of at least 16.2 days of life.
  Participants | 694
>= 1 pulmonary visit in study period [Count of Participants; unit: Participants] — To ensure the patient population was stable across study periods, we assessed patient characteristics including receipt of care in pulmonary clinics at Baseline Period. This is a baseline characteristic measured in the Baseline Period, not a study outcome.
  Participants | 42
Time smoked [Median (Inter-Quartile Range); unit: years] | 40.0 [30.0 to 45.0]
Cigarettes per day [Median (Inter-Quartile Range); unit: cigarettes per day] | 20.0 [20.0 to 30.0]
Current smoker [Count of Participants; unit: Participants] | 550
Former smoker (quit < 15 y ago) [Count of Participants; unit: Participants] | 554
Time since last smoked [Median (Inter-Quartile Range); unit: years] | 7.0 [3.9 to 10.7]
Insurance [Count of Participants; unit: Participants]
  Commercial | 337
  Government | 725
  Self-pay | 42
Patient portal use in preceding year [Count of Participants; unit: Participants] | 700
Telehealth primary care visit in preceding year [Count of Participants; unit: Participants] | 398
COVID-19 hospitalizations per day in Utah, median [Median (Inter-Quartile Range); unit: hospitalizations per participant] | 15.9 [0 to 25.9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Lung Cancer Screening (LCS) Care-Gap Closed
Description: The LCS care gap was considered closed if one or more of the following events occurred: (1) LDCT completion in the past year, (2) completion of another chest CT in the past year, or (3) SDM documentation in the past 3 years for eligible patients. To assess population care-gap closure levels at the end of each study period, we estimated the care-gap closure status for all patients who had primary care visits in the 12 months preceding the last day of the period. Using structured EHR data, SDM was considered documented if a clinician noted the need for LCS discussion was addressed, the patient declined screening, or LCS was not appropriate.
Time Frame: Through study completion, an average of 18 months for the intervention period and 12 months for the baseline period
Measure: Count of Participants; unit: Participants
Groups:
- Patients Eligible for LDCT Lung Cancer Screening: Patients aged 55-80 years who have smoked ≥30 pack-years and were a current smoker or quit smoking in the past 15 years.
Arm/Group | Patients Eligible for LDCT Lung Cancer Screening
Number analyzed (Participants) | 1255
Participants | 588

2. Other Pre Specified Outcome: Number of Participants Who Used the Intervention
Description: The number of participants who used the intervention was measured. The usage was measured through system logs and data from the enterprise data warehouse.
Time Frame: Through study completion, an average of 18 months for the intervention period
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Eligible for LDCT Lung Cancer Screening
Number analyzed (Participants) | 1255
Participants | 168

ADVERSE EVENTS:
Time Frame: The study period included 12 months baseline period and 18 months post-intervention implementation period.
Description: All-cause mortality in the preceding year was determined from the EHR data during the study period.
  Other adverse events were determined from the provider's and patient's reports.
Arm/Group | Patients Eligible for LDCT Lung Cancer Screening
All-Cause Mortality (participants affected / at risk) | 26/1255
Serious Adverse Events (participants affected / at risk) | 0/1255
Other Adverse Events (participants affected / at risk) | 0/1255

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT04498052/Prot_SAP_000.pdf